CLINICAL TRIAL: NCT06568159
Title: Patients with Coronary Artery Disease or At High Cardiovascular Risk: Measuring Compliance with Treatment for Obstructive Sleep Apnea Syndrome (OAM or CPAP)
Brief Title: Patients with Coronary Artery Disease or At High Cardiovascular Risk: Measuring Compliance with Treatment for Obstructive Sleep Apnea Syndrome
Acronym: PACOAM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0168
Record Dates: First submitted 2024-07-26; First posted 2024-08-23 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea; Coronary Disease; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Apnea, Obstructive; Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MAD group: * An oral and dental check-up will be carried out on the day of inclusion, and a sleep diary will be provided.
  * Compliance will be assessed after 6 months' wear.
  * As part of the research, specific questionnaires will be completed with the patient during a telephone interview after 6 months: assessment of compliance and quality of life.
- CPAP group: * An oral and dental check-up will be carried out on the day of inclusion.
  * Compliance will be assessed after 6 months' wear.
  * As part of the research, specific questionnaires will be completed with the patient during a telephone interview after 6 months: assessment of compliance and quality of life.

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder characterised by partial or total obstruction of the oro-pharyngeal carrefour during sleep. It is found in between 4% and 25% of the general population and in 40 to 80% of patients with cardiovascular diseases.

Continuous positive airway pressure (CPAP) is the standard treatment for OSA and its efficacy has already been demonstrated in this particular population. However, this treatment is not always accepted or sufficiently tolerated. The mandibular advancement device (MAD) is therefore an alternative treatment for OSA, validated by the French National Authority for Health and particularly relevant in this population because it is generally better tolerated. The aim of our study was to assess compliance, tolerance and usability of CPAP and MAD in patients with coronary artery disease and moderate (Apnea-Hypopnea Index AHI 15-30) to severe (AHI>30) OSA.

ELIGIBILITY:
Inclusion Criteria:

Target population: with coronary artery disease or at very high risk of coronary artery disease:

* Patients with coronary artery disease with or without co-morbidities (smoking, diabetes, hypertension, dyslipidaemia, renal insufficiency, overweight, emerging factors including anxiety-depression, shift workers, etc.).
* Hypertensive patients at high cardiovascular risk (target organ damage such as LVH or albuminuria)
* Diabetic patients at high cardiovascular risk
* Type of heart disease: ischaemic heart disease without clinically significant heart failure (NYHA II, III, IV) For the experimental group (MAD): patients with moderate or severe OSA with intolerance or refusal of CPAP and managed by MAD.

For the control group (CPAP): patients with moderate or severe OSA treated with CPAP.

Exclusion Criteria:

* Patients with heart failure not stabilised according to the investigator (NYHA IV)
* Severe psychiatric disorders
* Pregnant or breast-feeding women
* Opposition to participation after a period of reflection
* Not affiliated to a social security scheme,
* Persons under court protection,
* Persons under guardianship or curatorship
* Person taking part in another study with an exclusion period still in progress
* Inability to follow the patient during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged over 18, suffering from moderate to severe OSA and with CV pathology or at high risk of developing it.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Compliance with MAD and CPAP at 6 months (wearing time). | 6 months post-inclusion
  MAD compliance at 6 months (wearing time): a sleep diary will be given to the patient at the inclusion visit.
  CPAP compliance at 6 months: data transmitted by the CPAP device (sleep diary).

SECONDARY OUTCOMES:
Assessment of oral status | the day of inclusion
  plaque index : values from 0 to 3. A high score is a worse outcome.
Assessment of oral status | the day of inclusion
  mobility index : values from 1 to 4. A high score is a worse outcome.
Assessment of oral status | the day of inclusion
  bleeding index : values from 0 to 1 (100%). A high score is a worse outcome.
Assessment of tolerance and satisfaction with the device used reported by the patient at 6 months (duration of wear) | 6 months post-inclusion
  survey : values from 0 to 3. A high score is a better outcome.
Clinical parameters of OSA (objective) | 6 months post-inclusion
  ventilatory polygraphy or polysomnography
Assessment of quality of life | 6 months post-inclusion
  Survey WHOQOL Bref. Values : very poor, poor, neither poor nor good, good, very good.
Clinical parameters of OSA (subjective) | 6 months post-inclusion
  Survey. Values : light, moderate, significant

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de MONTPELLIER, Montpellier, France

IPD SHARING:
Plan to Share IPD: No